CLINICAL TRIAL: NCT02797912
Title: Nutritional Status and Pulmonary and Respiratory Muscle Function in Children and Young People With Cystic Fibrosis
Brief Title: LBM & Lung Function in Adolescents With CF
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: KCH16-074
Record Dates: First submitted 2016-06-08; First posted 2016-06-14 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
Keywords: pulmonary function; respiratory muscle function; body composition; exercise tolerance
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CF children and young people: Observational study involving clinical procedures: lung function testing, respiratory muscle strength testing, body composition analysis & exercise tolerance.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
In patients with cystic fibrosis (CF) the commonest cause of death is respiratory failure. Respiratory failure can have many causes. However, in patients with CF a major contributor is the impairment of the muscles required for breathing (respiratory muscles). Respiratory muscle impairment can result from poor nutrition. Lung function declines particularly during adolescence whilst body composition also changes at the same time. Thus, the investigators plan to study the relationship of nutrition and body composition to respiratory muscle strength and lung function in children and young people with CF aged between 12-18 years. The body mass index (BMI) is currently used in the clinical setting to measure nutritional status in CF. At King's College Hospital (KCH) there are portable devices to assess both respiratory muscle function and lung function. The research team will use a Bioelectrical Impedance Analysis (BIA) device to assess body composition, including BMI and lean body mass (LBM). The aim of the study is primarily to assess whether measurements of LBM impairment may better relate to poor lung function compared to BMI and secondly to examine whether lung and respiratory muscle function correlates with exercise tolerance.

DETAILED DESCRIPTION:
In patients with Cystic Fibrosis (CF) the commonest cause of death is respiratory failure. Respiratory failure can have many causes. However, in patients with CF a major contributor is the impairment of the muscles required for breathing (respiratory muscles). Respiratory muscle impairment can result from severe narrowing of the airways, poor nutrition, chronic infection and inflammation, lack of aerobic exercise and use of steroids (Dassios, 2015). The most rapid decline in lung function is seen during adolescence and coincides with a change in body composition (Loomba-Albrecht, 2009). The body mass index (BMI) is currently used in the clinical setting to quantify nutritional status in CF. However, measurements of the proportion of lean muscle, such as lean body mass (LBM), may better describe nutritional impairment in CF (Pedreira, 2005, Ionescu, 1998). LBM and BMI have been measured using dual x-ray absorptiometry (DXA) in children and young adults with CF showing a stronger association of LBM rather than BMI with pulmonary function especially in the undernourished adolescent (Sheikh, 2014). Assessment of respiratory muscle function and body composition has previously required specialised equipment, such as DXA, which is not readily available in many CF clinics. In addition, DXA involves radiation which may have unwanted side effects if used routinely for body composition monitoring. At King's College Hospital there are now, however, portable devices to assess both respiratory muscle function and body composition. The investigators will use a Bioelectrical Impedance Analysis (BIA) device to calculate body composition, including BMI and LBM. The aim of the study is primarily to assess whether LBM rather than BMI better predicts both pulmonary and respiratory muscle function using portable equipment that avoids use of avoidable radiation. Secondly, the research team aims to examine whether pulmonary and respiratory muscle function correlates to exercise capacity. These may yield useful information about targeting nutritional support and exercise to improve respiratory muscle and pulmonary function.

A cross-sectional study will be undertaken. Age, height, and weight will be recorded. Spirometry, impulse oscillometry and body plethysmography will be measured with a pneumotachograph based system (Jaeger Masterscreen PFT, Carefusion Ltd, Basingstoke UK) according to the American Thoracic Society and the European Respiratory Society guidelines. The highest value of forced vital capacity (FVC), forced expiratory volume in one second (FEV1), ratio of FEV1 to VC (FEV1/VC), forced expiratory flow between 25 and 75% of VC (FEF 25-75%), functional residual capacity (FRC), residual volume (RV), total lung capacity (TLC), respiratory system resistance at 5Hz and 20Hz (Rrs5, Rrs20) will be recorded following at least three technically acceptable measurements. Respiratory muscle function data will be obtained from the Micro RPM Respiratory Muscle Analyser (CareFusion, San Diego, California, USA): maximum inspiratory pressure (MIP), maximum expiratory pressure (MEP), sniff nasal inspiratory pressure (SNIP), maximum relaxation rate (MRR), time constant of relaxation (τ, tau), and maximum rate of pressure development (MRPD). A respiratory health questionnaire will be completed. Body composition information will be obtained with the Inbody S10 Body Composition Analyzer (Inbody Ltd, Cerritos, California, USA): Body mass index (BMI), BMI-z scores, fat free mass (FFM), segmental lean mass (LM) [LM-right arm (LMRA), LM-left arm (LMLA), LM-trunk (LMTR), LM-right leg (LMRL), LM-left leg (LMLL)], visceral fat area (VFA), body cell mass (BCM). A field test to assess exercise tolerance test will be performed and the level of habitual activity will be assessed using a questionnaire. Information will be collected on genetic mutations, chronic infection status, use of systemic corticosteroids, and co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* Ages 12-19

Exclusion Criteria:

* Acute illness or hospitalisation that would render the participants unable to undertake the assessment, including pulmonary exacerbation in past 2-weeks,

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young people with confirmed CF, between 12 years and 18 will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Association between body mass index (BMI) & lean body mass (LBM) with pulmonary & respiratory muscle function | 4 months

SECONDARY OUTCOMES:
Association between exercise tolerance and pulmonary & respiratory muscle function | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation School, London, United Kingdom

REFERENCES:
- [Background] Dassios T. Determinants of respiratory pump function in patients with cystic fibrosis. Paediatr Respir Rev. 2015 Jan;16(1):75-9. doi: 10.1016/j.prrv.2014.01.001. Epub 2014 Jan 28. PMID 24661942
- [Background] Loomba-Albrecht LA, Styne DM. Effect of puberty on body composition. Curr Opin Endocrinol Diabetes Obes. 2009 Feb;16(1):10-5. doi: 10.1097/med.0b013e328320d54c. PMID 19115520
- [Background] Pedreira CC, Robert RG, Dalton V, Oliver MR, Carlin JB, Robinson P, Cameron FJ. Association of body composition and lung function in children with cystic fibrosis. Pediatr Pulmonol. 2005 Mar;39(3):276-80. doi: 10.1002/ppul.20162. PMID 15668934
- [Background] Ionescu AA, Chatham K, Davies CA, Nixon LS, Enright S, Shale DJ. Inspiratory muscle function and body composition in cystic fibrosis. Am J Respir Crit Care Med. 1998 Oct;158(4):1271-6. doi: 10.1164/ajrccm.158.4.9710079. PMID 9769291
- [Background] Sheikh S, Zemel BS, Stallings VA, Rubenstein RC, Kelly A. Body composition and pulmonary function in cystic fibrosis. Front Pediatr. 2014 Apr 15;2:33. doi: 10.3389/fped.2014.00033. eCollection 2014. PMID 24783186